CLINICAL TRIAL: NCT03845517
Title: A PHASE 2B, DOUBLE-BLIND, RANDOMIZED, PLACEBO-CONTROLLED, MULTICENTER, DOSE-RANGING STUDY TO EVALUATE THE EFFICACY AND SAFETY PROFILE OF PF-06700841 IN PARTICIPANTS WITH ACTIVE SYSTEMIC LUPUS ERYTHEMATOSUS (SLE)
Brief Title: A DOSE-RANGING STUDY TO EVALUATE EFFICACY AND SAFETY OF PF-06700841 IN SYSTEMIC LUPUS ERYTHEMATOSUS (SLE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B7931028; 2018-004175-12 (EudraCT Number)
Record Dates: First submitted 2019-02-15; First posted 2019-02-19 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — PF-06700841

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- PF-06700841 15 mg (Experimental): PF-06700841 15 mg
  Interventions: Drug: PF-06700841 15 mg
- PF-06700841 30 mg (Experimental): PF-06700841 30 mg
  Interventions: Drug: PF-06700841 30 mg
- PF-06700841 45 mg (Experimental): PF-06700841 45 mg
  Interventions: Drug: PF-06700841 45 mg

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: PF-06700841 15 mg — PF-06700841 15 mg
  Arms: PF-06700841 15 mg
Drug: PF-06700841 30 mg — PF-06700841 30 mg
  Arms: PF-06700841 30 mg
Drug: PF-06700841 45 mg — PF-06700841 45 mg
  Arms: PF-06700841 45 mg

SUMMARY:
Assessment of PF-06700841 in participants with moderate to severe active, generalized Systemic Lupus Erythematosus (SLE) that have inadequate response to standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female subjects between ≥18 and ≤75 years of age inclusive.
* Diagnosis of moderate to severe active Lupus.
* Receiving a stable dose of methotrexate, azathioprine, leflunomide, mizoribine, mycophenolate/mycophenolic acid, anti-malarials or corticosteroids.

Exclusion Criteria:

* Active renal lupus
* Severe active central nervous system (CNS) lupus
* Have cancer or a history of cancer within 5 years of screening.
* Have a history of thrombosis (venous or arterial) or other vascular complications within the last 6 months, or any history of either recurrent thrombosis or a pulmonary embolus.
* Active bacterial, viral, fungal, mycobacterial or other infections
* Psychiatric condition including recent or active suicidal ideation or behavior
* Have active fibromyalgia/myofascial/chronic pain.
* Pregnant female subjects; breastfeeding female subjects; females subjects planning to become pregnant during the study; fertile male subjects and WOCBP who are unwilling or unable to use a highly effective method of contraception.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (162):
- United States (54):
  - UAB Department of Medicine Clinical Research Enterprise, Birmingham, Alabama
  - The Kirklin Clinic, Birmingham, Alabama
  - UAB Hospital Department of Pharmacy, Birmingham, Alabama
  - UAB Hospital-Clinical Research Unit (CRU), Birmingham, Alabama
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - St. Joseph Heritage Healthcare, Fullerton, California
  - Advanced Medical Research, LLC, La Palma, California
  - Arthritis and Osteoporosis Medical Center, La Palma, California
  - Desert Medical Advances, Palm Desert, California
  - East Bay Rheumatology Medical Group, Inc., San Leandro, California
  - Millennium Clinical Trials, Thousand Oaks, California
  - Inland Rheumatology and Osteoporosis Medical Group, Upland, California
  - Inland Rheumatology Clinical Trials, Inc., Upland, California
  - New England Research Associates, LLC, Bridgeport, Connecticut
  - New England Research Associates, Bridgeport, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Clinical Research of West Florida, Clearwater, Florida
  - Private Practice of Robert W. Levin, Clearwater, Florida
  - SIMEDHealth, LLC Attn: Rheumatology, Gainesville, Florida
  - SIMEDHealth, LLC, Gainesville, Florida
  - Omega Research MetroWest, LLC, Orlando, Florida
  - Akumin, Inc, Palm Harbor, Florida
  - Akumin Inc, St. Petersburg, Florida
  - West Broward Rheumatology Associates, Inc, Tamarac, Florida
  - Akumin Inc., Tampa, Florida
  - Rose Radiology dba Akumin Inc., Tampa, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - AdventHealth Tampa, Tampa, Florida
  - Jefrey D. Lieberman, M.D., P.C., Decatur, Georgia
  - Atlanta Research Center for Rheumatology, Marietta, Georgia
  - Institute of Arthritis Research, Idaho Falls, Idaho
  - Investigational Drug Services University of Kansas Hospital, Kansas City, Kansas
  - The University of Kansas Hospital, Kansas City, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - Ochsner Clinic Foundation, Baton Rouge, Baton Rouge, Louisiana
  - University of Michigan Brighton Center for Specialty Care, Brighton, Michigan
  - Innovative health Research, Las Vegas, Nevada
  - NYU Langone Ambulatory Care Brooklyn Heights, Brooklyn, New York
  - St. Lawrence Health System, Canton, New York
  - Feinstein Institute for Medical Research, Manhasset, New York
  - Northshore University Hospital, Manhasset, New York
  - Columbia University Medical Center., New York, New York
  - Irving Institute for Clinical and Transitional Research, New York, New York
  - St. Lawrence Health System, Potsdam, New York
  - Joint and Muscle Research Institute, Charlotte, North Carolina
  - Arthritis & Rheumatology Center of Oklahoma PLLC, Oklahoma City, Oklahoma
  - West Tennessee Research Institute, Jackson, Tennessee
  - Gupta, Ramesh C MD, Memphis, Tennessee
  - Tekton Research, Austin, Texas
  - Accurate Clinical Management, LLC, Baytown, Texas
  - Rheumatic Disease Clinical Research Center, LLC, Houston, Texas
  - Accurate Clinical Research, Houston, Texas
  - Arthritis Clinic of Central Texas, San Marcos, Texas
  - Arthritis Northwest, PLLC, Spokane, Washington
- Centro de Investigaciones Medicas Tucuman, San Miguel de Tucumán, Tucumán Province, Argentina
- Australia (2):
  - Optimus Clinical Research, Kogarah, New South Wales
  - Emeritus Research, Camberwell, Victoria
- Belgium (2):
  - UZ Leuven, Leuven
  - Ziekenhuisnetwerk Antwerpen Jan Palfijn (ZNA Jan Palfijn), Merksem
- Bulgaria (5):
  - DCC Sveti Georgi EOOD, Plovdiv
  - MHAT Plovdiv AD, Plovdiv
  - Umhat Kanev Ad, Rousse
  - UMHAT "Sv.Ivan Rilski" EAD, Sofia
  - UMHAT "Sv. Ivan Rilski" EAD, Sofia
- Canada (2):
  - Centre intégré de santé et de services sociaux du Bas-Saint-Laurent, Rimouski, Quebec
  - Centre de Recherche Musculo-Squelettique, Trois-Rivières, Quebec
- China (7):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Peking Union Medical College Hospital, Beijing
  - Ruijin Hospital- Shanghai Jiaotong University School of Medicine, Shanghai
  - Fudan University Hua Shan Hospital, Shanghai
- Colombia (5):
  - Hospital Pablo Tobon Uribe, Medellín, Antioquia
  - Centro Integral de Reumatología del Caribe S.A.S - CIRCARIBE S.A.S, Barranquilla, Atlántico
  - Bluecare Salud S.A.S Sede Centro Médico Integral Chicó MedPlus CRI, Bogota, Cundinamarca
  - Centro de Investigación en Reumatología y Especialidades Médicas SAS - CIREEM SAS, Bogotá, Cundinamarca
  - Medicity S.A.S., Bucaramanga, Santander Department
- Czechia (3):
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Nemocnicni lekarna VFN, Prague
  - Revmatologicky ustav, Prague
- France (3):
  - Hôpital Pitié Salpêtrière, Centre des Maladies Auto-immunes, Paris
  - Hôpital Cochin, Paris
  - CHU de Bordeaux, Groupe Hospitalier Sud, Hôpital Haut Lévèque, Pessac
- Germany (2):
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Schleswig Holstein - Campus Lübeck, Lübeck
- Greece (3):
  - University General Hospital of Heraklion, Heraklion, Crete
  - Laiko General Hospital, University of Athens, Athens
  - University Hospital ATTIKON, Haidari
- Tuen Mun Hospital, Hong Kong, Hong Kong
- Hungary (3):
  - Qualiclinic Kft., Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Békés Vármegyei Központi Kórház, Gyula
- Fondazione IRCCS Policlinico S.Matteo, Pavia, Italy
- Japan (9):
  - National Hospital Organization Asahikawa Medical Center, Asahikawa, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Tohoku University Hospital, Sendai, Miyagi
  - Sasebo Chuo Hospital, Sasebo, Nagasaki
  - Shinkenko clinic, Naha, Okinawa
  - St. Luke's International Hospital, Chuo-ku, Tokyo
  - National Hospital Organization Chiba-East Hospital, Chiba
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Hiroshima University Hospital, Hiroshima
- Mexico (9):
  - CITER Centro de Investigación y Tratamiento de las Enfermedades Reumáticas S.A. de C.V., Mexico City, Cuauhtémoc
  - Morales Vargas Centro de Investigación S.C., León, Guanajuato
  - Investigación Biomédica para el Desarrollo de Fármacos S.A. de C.V, Guadalajara, Jalisco
  - Investigación Biomédica para el Desarrollo de Fármacos S.A. de C.V, Zapopan, Jalisco
  - Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Tlalpan
  - Centro Peninsular de Investigación Clínica S.C.P., Mérida, Yucatán
  - Investigación y Biomedicina de Chihuahua, Sociedad Civil, Chihuahua City
  - Investigación Biomédica para el Desarrollo de Fármacos S.A. de C.V, Guadalajara
  - CINTRE Centro de Investigación y Tratamiento Reumatológico S.C., Mexico City
- Poland (8):
  - Centrum Wsparcia Badan Klinicznych, Warsaw, Masovian Voivodeship
  - Stanislaw Sierakowski Centrum Miriada, Bialystok
  - Szpital Biziela, Bydgoszcz
  - Zespol Poradni Specjalistycznych Reumed, Onyksowa Filia nr 2, Lublin
  - NZOZ "Lecznica Mak-Med" s.c., Nadarzyn
  - Centrum Medyczne MEDENS S.C. Grupowa Praktyka Lekarska, Sosnowiec
  - Narodowy Instytutu Geriatrii, Reumatologii i Rehabilitacji, Warsaw
  - Mazowieckie Centrum Reumatologii i Osteoporozy M. Przygodzka Spolka jawna, Warsaw
- Portugal (4):
  - Hospital Garcia de Orta, E.P.E, Almada
  - Hospital Professor Doutor Fernando da Fonseca, E.P.E, Amadora
  - Unidade Local de Saude do Alto Minho, E.P.E., Ponte de Lima
  - Centro Hospitalar Universitario do Porto, E.P.E, Porto
- Romania (4):
  - SC Centrul Medical de Diagnostic si Tratament Ambulator Neomed SRL, Brasov, JUD. Brasov
  - Spitalul Clinic Judetean de Urgenta Cluj-Napoca, Cluj-Napoca, JUD. CLUJ
  - S.C. Euroclinic Hospital S.A, Bucharest, Sector 1
  - Spitalul Clinic Sf. Maria, Bucharest
- Serbia (4):
  - Institut za Reumatologiju, Belgrade
  - Klinicki Centar Srbije, Klinika za alergologiju i imunologiju, Belgrade
  - Vojnomedicinska akademija, Klinika za reumatologiju, Belgrade
  - Institut Niska Banja, Klinika za Reumatologiju, Niška Banja
- South Korea (3):
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seocho-gu, Seoul
  - Kyungpook National University Hospital (KNUH), Daegu
- Spain (6):
  - Hospital do Meixoeiro, Vigo, Pontevedra
  - Complexo Hospitalario Universitario A Coruna, A Coruña
  - Hospital Germans Trias i Pujol, Badalona
  - Clinica Sagrada Familia, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Quiron Infanta Luisa, Seville
- Taiwan (8):
  - China Medical University Hospital, Taichung, Taiwan (r.o.c)
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital Linkou Branch, Taoyuan
- Ukraine (9):
  - State Institution National Scientific Center "M.D. Strazhesko Institute of Cardiology" of National, Kyiv
  - State Institution National Scientific Center "M.D. Strazhesko Institute of Cardiology", Kyiv
  - Communal non-profitable enterprise "Lviv City Clinical Hospital #4", Lviv
  - Multifield Medical Center of Odesa National Medical University, Odesa
  - Multifield Medical Center of Odessa National Medical University, Odesa
  - CNPE "Odesa Regional Clinical Hospital" of Odesa Regional Council, Odesa
  - CNPE "Ternopil University Hospital" of Ternopil regional council, Department of Rheumatology, Ternopil
  - Zakarpattia Regional Clinical Hospital n.a. A. Novak, Uzhhorod
  - CNPE "Vinnytsya regional Clinical Hospital named after N.I.Pirogov Vinnytsia Regional Council", Vinnytsia
- United Kingdom (4):
  - Southampton General Hospital, Southampton, Hampshire
  - Doncaster Royal Infirmary, Doncaster and Bassetlaw Teaching Hospitals NHS Foundation Trust, Doncaster
  - The Leeds Teaching Hospitals NHS Trust, Chapel Allerton Hospital, Leeds
  - Guy's and St Thomas' NHS Foundation Trust Guy's Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7931028

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 350 participants with active systemic lupus erythematosus (SLE) were enrolled and randomized in the study.
Groups:
- Placebo: Participants were randomized to receive placebo matched to PF-06700841 once daily (QD) for 52 weeks. Participants were followed up for 4 weeks after last dose.
- PF-06700841 15 mg: Participants were randomized to receive PF-06700841 15 milligrams (mg) tablets orally QD for 52 weeks. Participants were followed up for 4 weeks after last dose.
- PF-06700841 30 mg: Participants were randomized to receive PF-06700841 30 mg tablets orally QD for 52 weeks. Participants were followed up for 4 weeks after last dose.
- PF-06700841 45 mg: Participants were randomized to receive PF-06700841 45 mg tablets orally QD for 52 weeks. Participants were followed up for 4 weeks after last dose.
Period: Treatment Period (52 Weeks)
Arm/Group | Placebo | PF-06700841 15 mg | PF-06700841 30 mg | PF-06700841 45 mg
Started | 100 | 50 | 101 | 99
Completed | 68 | 36 | 78 | 71
Not Completed | 32 | 14 | 23 | 28
Not completed — Adverse Event | 12 | 7 | 10 | 17
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 8 | 1 | 3 | 4
Not completed — Lost to Follow-up | 2 | 0 | 1 | 0
Not completed — Non-compliance with study drug | 1 | 0 | 0 | 0
Not completed — Physician's decision | 0 | 0 | 1 | 0
Not completed — Site Terminated by Sponsor | 2 | 0 | 0 | 0
Not completed — Other | 2 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 4 | 6 | 6 | 5
Period: Follow-up Period (4 Weeks)
Arm/Group | Placebo | PF-06700841 15 mg | PF-06700841 30 mg | PF-06700841 45 mg
Started | 100 (Participants who started treatment phase entered in follow-up phase.) | 50 (Participants who started treatment phase entered in follow-up phase.) | 101 (Participants who started treatment phase entered in follow-up phase.) | 99 (Participants who started treatment phase entered in follow-up phase.)
Completed | 89 | 42 | 89 | 92
Not Completed | 11 | 8 | 12 | 7
Not completed — Adverse Event | 4 | 2 | 0 | 2
Not completed — Death | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 2 | 1 | 2 | 0
Not completed — Physician's decision | 0 | 0 | 1 | 1
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 1
Not completed — Other | 1 | 0 | 1 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 5 | 7 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who were randomly assigned to study intervention and who took at least 1 dose of study intervention.
Groups:
- Placebo: Participants were randomized to receive placebo matched to PF-06700841 QD for 52 weeks. Participants were followed up for 4 weeks after last dose.
- PF-06700841 15 mg: Participants were randomized to receive PF-06700841 15 mg tablets orally QD for 52 weeks. Participants were followed up for 4 weeks after last dose.
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-06700841 15 mg | PF-06700841 30 mg | PF-06700841 45 mg | Total
Number analyzed (Participants) | 100 | 50 | 101 | 99 | 350
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.5 (9.60) | 41.5 (11.79) | 42.8 (12.71) | 41.0 (11.47) | 42.0 (11.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 45 | 97 | 91 | 327
  Male | 6 | 5 | 4 | 8 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 17 | 34 | 35 | 115
  Not Hispanic or Latino | 71 | 32 | 67 | 62 | 232
  Unknown or Not Reported | 0 | 1 | 0 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 7 | 2 | 11
  Asian | 14 | 9 | 11 | 13 | 47
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 4 | 6 | 7 | 23
  White | 71 | 31 | 69 | 68 | 239
  More than one race | 2 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 5 | 6 | 8 | 9 | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving SLE Responder Index (SRI) Change of 4 (SRI-4) at Week 52
Description: SRI-4 components included Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K), British Isles Lupus Assessment Group (BILAG) 2004 and Physician's Global Assessment (PhGA). Participants were classified as SRI-4 responders, if they met all of the following criteria compared with baseline: 1) greater than or equal to (>=) 4 point reduction in SLEDAI-2K score; 2) no new BILAG A organ domain score or 2 new BILAG B organ domain scores; 3) no worsening (less than [<] 0.3 point increase) in PhGA score. SLEDAI-2K: assesses improvement in disease activity (range: 0 to 105; higher score = higher severity). BILAG: assesses disease extent, severity in individual organ system (range: A [severe] to E [no disease]; higher score = less severity). PhGA: assesses worsening in participant's general health status (range: 0 [none] to 3 [severe]; higher score = higher severity).
Time Frame: Week 52
Population: Full analysis set (FAS) included all participants randomly assigned to study intervention and have received at least 1 dose of study intervention. Here "Number of Participants Analyzed" signifies participants at Week 52 with Non-Responder Imputation (NRI) and Last Observation Carried Forward from Week 48 (LOCF48) applied.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-06700841 15 mg | PF-06700841 30 mg | PF-06700841 45 mg
Number analyzed (Participants) | 96 | 47 | 99 | 92
Percentage of participants | 64.6 [54.5 to 74.7] | 57.4 [42.2 to 72.6] | 69.7 [60.1 to 79.3] | 66.3 [56.1 to 76.5]
Statistical Analysis 1: Comparison: Placebo vs PF-06700841 15 mg; Test type: Superiority; p = 0.8076, Cochran-Mantel-Haenszel — One sided p-value; Risk Difference (RD) = -7.5, 95% CI 2-sided [-24.5 to 9.5]
Statistical Analysis 2: Comparison: Placebo vs PF-06700841 30 mg; Test type: Superiority; p = 0.2189, Cochran-Mantel-Haenszel — One sided p-value; Risk Difference (RD) = 5.2, 95% CI 2-sided [-7.9 to 18.3]
Statistical Analysis 3: Comparison: Placebo vs PF-06700841 45 mg; Test type: Superiority; p = 0.4010, Cochran-Mantel-Haenszel — One sided p-value; Risk Difference (RD) = 1.7, 95% CI 2-sided [-11.8 to 15.3]

2. Secondary Outcome: Percentage of Participants Achieving British Isles Lupus Assessment Group-Based Composite Lupus Assessment (BICLA) at Week 52
Description: BICLA included: BILAG-2004, SLEDAI-2K and PhGA. Participants were classified as responders, if they met all the following criteria: BILAG-2004 improvement (all A scores at baseline improved to B/C/D and all B scores improved to C or D); no worsening in disease activity (no new BILAG-2004 A scores or =<1 new B score); no worsening of total SLEDAI-2K score; no significant deterioration (<10 percent [%] worsening) in analogue PhGA. SLEDAI-2K: assesses improvement in disease activity (range: 0 to 105; higher score = higher severity). BILAG: assesses disease extent, severity in individual organ system (range: A [severe] to E [no disease]; higher score = less severity). PhGA: assesses worsening in participant's general health status (range: 0 [none] to 3 [severe]; higher score = higher severity).
Time Frame: Week 52
Population: FAS included all participants randomly assigned to study intervention and have received at least 1 dose of study intervention. Here "Number of Participants Analyzed" signifies participants at Week 52 with NRI and LOCF48 applied.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-06700841 15 mg | PF-06700841 30 mg | PF-06700841 45 mg
Number analyzed (Participants) | 96 | 47 | 99 | 92
Percentage of participants | 43.8 [33.3 to 54.2] | 42.6 [27.4 to 57.8] | 52.5 [42.2 to 62.9] | 53.3 [42.5 to 64.0]
Statistical Analysis 1: Comparison: Placebo vs PF-06700841 15 mg; Test type: Superiority; p = 0.5950, Cochran-Mantel-Haenszel — One sided p-value; Risk Difference (RD) = -2.1, 95% CI 2-sided [-19.1 to 14.9]
Statistical Analysis 2: Comparison: Placebo vs PF-06700841 30 mg; Test type: Superiority; p = 0.1125, Cochran-Mantel-Haenszel — One sided p-value; Risk Difference (RD) = 8.6, 95% CI 2-sided [-5.3 to 22.6]
Statistical Analysis 3: Comparison: Placebo vs PF-06700841 45 mg; Test type: Superiority; p = 0.0891, Cochran-Mantel-Haenszel — One sided p-value; Risk Difference (RD) = 9.6, 95% CI 2-sided [-4.4 to 23.6]

3. Secondary Outcome: Percentage of Participants Achieving Lupus Low Disease Activity State (LLDAS) at Week 52
Description: LLDAS was defined as SLE disease activity index (SLEDAI-2k <=4, with no activity in major organ systems [renal, central nervous system, cardiopulmonary, vasculitis, fever]) and no haemolytic anaemia or gastrointestinal activity; no new lupus disease activity compared with the previous assessment; a Safety of Estrogens in Lupus Erythematosus National Assessment (SELENA)-SLEDAI PhGA (scale 0-3; higher scores = higher severity) <=1; a current prednisolone (or equivalent) dose <=7.5 milligram per day (mg/daily); and well tolerated standard maintenance doses of immunosuppressive drugs and approved biological agents.
Time Frame: Week 52
Population: FAS included all participants randomly assigned to study intervention and have received at least 1 dose of study intervention. Here "Number of Participants Analyzed" signifies participants at Week 52 with NRI applied.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-06700841 15 mg | PF-06700841 30 mg | PF-06700841 45 mg
Number analyzed (Participants) | 93 | 47 | 97 | 88
Percentage of participants | 22.6 [13.5 to 31.6] | 21.3 [8.5 to 34.0] | 35.1 [25.0 to 45.1] | 34.1 [23.6 to 44.6]

4. Secondary Outcome: Percentage of Participants Achieving a Reduction in Prednisone (or Equivalent) Dose to <=7.5 mg/Day and Sustained for 12 Weeks Prior to Week 52 in Participants on Prednisone >7.5 mg/Day (or Equivalent) at Baseline
Description: In this outcome measure data is reported for participants who achieved a reduction in prednisone (or equivalent) dose to <=7.5 mg/day and sustained for 12 Weeks prior at Week 52 and they also sustained this dose reduction for 12 weeks prior to Week 52 (Week 40 to Week 52).
Time Frame: Week 52 for achieving reduction in dose along with Week 40 to Week 52 for sustained dosing
Population: FAS included all participants randomly assigned to study intervention and have received at least 1 dose of study intervention. Number of participants in FAS with baseline Prednisone or equivalent >7.5 mg/day were analyzed. Here, "Number of Participants Analyzed" signifies participants at Week 52 with NRI applied.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-06700841 15 mg | PF-06700841 30 mg | PF-06700841 45 mg
Number analyzed (Participants) | 53 | 33 | 46 | 43
Percentage of participants | 26.4 [13.6 to 39.2] | 36.4 [18.4 to 54.3] | 37.0 [21.9 to 52.0] | 41.9 [26.0 to 57.8]

5. Secondary Outcome: Percentage of Participants Achieving a SRI-4 Response With Prednisone Dose Reduced to <=7.5 mg/Day and Sustained for 12 Weeks at Week 52 in Participants on Prednisone >7.5 mg/Day (or Equivalent) at Baseline
Description: In this outcome measure data is reported for participants who achieved a reduction in SRI-4 response with prednisone dose reduced to <=7.5 mg/day and sustained for 12 weeks at Week 52.
Time Frame: 12 Weeks prior at Week 52 (Week 40 to Week 52)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-06700841 15 mg | PF-06700841 30 mg | PF-06700841 45 mg
Number analyzed (Participants) | 53 | 33 | 46 | 43
Percentage of participants | 20.8 [8.9 to 32.6] | 30.3 [13.1 to 47.5] | 32.6 [18.0 to 47.2] | 32.6 [17.4 to 47.7]

6. Secondary Outcome: Percentage of Participants With >= 50% Reduction in Cutaneous Lupus Erythematosus Disease Area and Severity Index Activity (CLASI-A) Score at Week 52 in Participants With Baseline CLASI-A Score >=10
Description: CLASI is an validated measurement instrument for lupus erythematosus developed for use in clinical studies that consists of separate scores for the activity of the disease (CLASI-A). The CLASI activity score is calculated on the basis of erythema, scale/hyperkeratosis, mucous membrane involvement, acute hair loss and non-scarring alopecia. The CLASI activity score ranges from 0-70, with higher scores indicating more severe skin disease. Severity categories based on the CLASI activity score are as follows: mild (0-9), moderate (10-20), and severe (21-70).
Time Frame: Week 52
Population: FAS included all participants randomly assigned to study intervention and have received at least 1 dose of study intervention. Number of participants in FAS with baseline CLASI-A score >= 10 were analyzed. Here, "Number of Participants Analyzed" signifies participants at Week 52 with NRI applied.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-06700841 15 mg | PF-06700841 30 mg | PF-06700841 45 mg
Number analyzed (Participants) | 23 | 12 | 27 | 16
Percentage of participants | 73.9 [53.8 to 94.0] | 58.3 [26.3 to 90.4] | 77.8 [60.2 to 95.3] | 56.3 [28.8 to 83.7]

7. Secondary Outcome: Change From Baseline in Total Scores of Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) at Week 52
Description: The FACIT-F Scale is a participant completed questionnaire consisting of 13 items that assess fatigue. Participants responded to each item on a 5-point scale based on their experience of fatigue during the past 7 days (0 = not at all; 1 = a little bit; 2 =somewhat; 3 = quite a bit; 4 = very much). Instrument scoring yielded a range from 0 to 52 (negatively worded items were reversed during analysis), with higher scores representing better participant status (less fatigue).
Time Frame: Baseline, Week 52
Population: FAS included all participants randomly assigned to study intervention and have received at least 1 dose of study intervention. Here, "Number of Participants Analyzed" signifies participants evaluable with observed data at Week 52.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo | PF-06700841 15 mg | PF-06700841 30 mg | PF-06700841 45 mg
Number analyzed (Participants) | 66 | 36 | 75 | 64
Units on a scale | 4.6 [2.5 to 6.6] | 7.4 [4.5 to 10.2] | 5.8 [3.8 to 7.8] | 7.6 [5.5 to 9.7]

8. Secondary Outcome: Change From Baseline in Physical Health Domain Scores of Lupus Quality of Life (LupusQoL) at Week 52
Description: The LupusQoL questionnaire is a validated questionnaire used to evaluate SLE -specific concepts of SLE as reported by participants. It consists of 34 items in 8 different domains: physical health, emotional health, body image, pain, planning, fatigue, intimate relationship, and burden to others; measured on a 5-point scale ranging from 0 (not at all) to 4 (very much). The individual domain scores are transformed to a 0 to 100 scale wherein higher scores indicate better quality of life. Physical health domain score of LupusQoL had score range from 0 to 100, where higher scores = better quality of life.
Time Frame: Baseline, Week 52
Population: FAS included all participants randomly assigned to study intervention and have received at least 1 dose of study intervention. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure with observed data at the specified visit.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo | PF-06700841 15 mg | PF-06700841 30 mg | PF-06700841 45 mg
Number analyzed (Participants) | 66 | 36 | 75 | 64
Units on a scale | 11.585 [7.475 to 15.695] | 10.892 [5.241 to 16.544] | 12.371 [8.464 to 16.278] | 14.875 [10.748 to 19.002]

9. Secondary Outcome: Change From Baseline in Emotional Health Domain Scores of LupusQoL at Week 52
Description: The LupusQoL questionnaire is a validated questionnaire used to evaluate SLE -specific concepts of SLE as reported by participants. It consists of 34 items in 8 different domains: physical health, emotional health, body image, pain, planning, fatigue, intimate relationship, and burden to others measured on a 5-point scale ranging from 0 (not at all) to 4 (very much). The individual domain scores are transformed to a 0 to 100 scale wherein higher scores indicate better quality of life. Emotional health domain score of LupusQoL had score range from 0 to 100, where higher scores = better quality of life.
Time Frame: Baseline, Week 52
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo | PF-06700841 15 mg | PF-06700841 30 mg | PF-06700841 45 mg
Number analyzed (Participants) | 66 | 36 | 75 | 64
Units on a scale | 8.113 [4.132 to 12.093] | 10.469 [4.968 to 15.969] | 7.547 [3.749 to 11.346] | 11.823 [7.806 to 15.840]

10. Secondary Outcome: Change From Baseline in Body Image Domain Scores of LupusQoL at Week 52
Description: The LupusQoL questionnaire is a validated questionnaire used to evaluate SLE -specific concepts of SLE as reported by participants. It consists of 34 items in 8 different domains: physical health, emotional health, body image, pain, planning, fatigue, intimate relationship, and burden to others measured on a 5-point scale ranging from 0 (not at all) to 4 (very much). The individual domain scores are transformed to a 0 to 100 scale wherein higher scores indicate better quality of life. Body image domain score of LupusQoL had score range from 0 to 100, where higher scores = better quality of life.
Time Frame: Baseline, Week 52
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo | PF-06700841 15 mg | PF-06700841 30 mg | PF-06700841 45 mg
Number analyzed (Participants) | 62 | 32 | 66 | 50
Units on a scale | 9.207 [4.352 to 14.062] | 10.935 [4.070 to 17.799] | 8.169 [3.448 to 12.890] | 15.599 [10.355 to 20.843]

11. Secondary Outcome: Change From Baseline in Pain Domain Scores of LupusQoL at Week 52
Description: The LupusQoL questionnaire is a validated questionnaire used to evaluate SLE -specific concepts of SLE as reported by participants. It consists of 34 items in 8 different domains: physical health, emotional health, body image, pain, planning, fatigue, intimate relationship, and burden to others measured on a 5-point scale ranging from 0 (not at all) to 4 (very much). The individual domain scores are transformed to a 0 to 100 scale wherein higher scores indicate better quality of life. Pain domain score of LupusQoL had score range from 0 to 100, where higher scores = better quality of life.
Time Frame: Baseline, Week 52
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo | PF-06700841 15 mg | PF-06700841 30 mg | PF-06700841 45 mg
Number analyzed (Participants) | 66 | 36 | 75 | 64
Units on a scale | 15.065 [10.470 to 19.659] | 15.480 [9.132 to 21.828] | 16.855 [12.488 to 21.223] | 24.418 [19.790 to 29.047]

12. Secondary Outcome: Change From Baseline in Planning Domain Scores of LupusQoL at Week 52
Description: The LupusQoL questionnaire is a validated questionnaire used to evaluate SLE -specific concepts of SLE as reported by participants. It consists of 34 items in 8 different domains: physical health, emotional health, body image, pain, planning, fatigue, intimate relationship, and burden to others measured on a 5-point scale ranging from 0 (not at all) to 4 (very much). The individual domain scores are transformed to a 0 to 100 scale wherein higher scores indicate better quality of life. Planning domain score of LupusQoL had score range from 0 to 100, where higher scores = better quality of life.
Time Frame: Baseline, Week 52
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo | PF-06700841 15 mg | PF-06700841 30 mg | PF-06700841 45 mg
Number analyzed (Participants) | 66 | 36 | 75 | 64
Units on a scale | 14.168 [9.423 to 18.912] | 12.013 [5.487 to 18.538] | 10.335 [5.826 to 14.843] | 20.310 [15.523 to 25.097]

13. Secondary Outcome: Change From Baseline in Fatigue Domain Scores of LupusQoL at Week 52
Description: The LupusQoL questionnaire is a validated questionnaire used to evaluate SLE -specific concepts of SLE as reported by participants. It consists of 34 items in 8 different domains: physical health, emotional health, body image, pain, planning, fatigue, intimate relationship, and burden to others measured on a 5-point scale ranging from 0 (not at all) to 4 (very much). The individual domain scores are transformed to a 0 to 100 scale wherein higher scores indicate better quality of life. Fatigue domain score of LupusQoL had score range from 0 to 100, where higher scores = better quality of life.
Time Frame: Baseline, Week 52
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo | PF-06700841 15 mg | PF-06700841 30 mg | PF-06700841 45 mg
Number analyzed (Participants) | 66 | 36 | 75 | 64
Units on a scale | 10.317 [5.951 to 14.683] | 11.893 [5.892 to 17.894] | 11.701 [7.550 to 15.853] | 16.443 [12.036 to 20.850]

14. Secondary Outcome: Change From Baseline in Intimate Relationship Domain Scores of LupusQoL at Week 52
Description: The LupusQoL questionnaire is a validated questionnaire used to evaluate SLE -specific concepts of SLE as reported by participants. It consists of 34 items in 8 different domains: physical health, emotional health, body image, pain, planning, fatigue, intimate relationship, and burden to others measured on a 5-point scale ranging from 0 (not at all) to 4 (very much). The individual domain scores are transformed to a 0 to 100 scale wherein higher scores indicate better quality of life. Intimate relationship domain score of LupusQoL had score range from 0 to 100, where higher scores = better quality of life.
Time Frame: Baseline, Week 52
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo | PF-06700841 15 mg | PF-06700841 30 mg | PF-06700841 45 mg
Number analyzed (Participants) | 56 | 25 | 59 | 42
Units on a scale | 12.430 [6.842 to 18.019] | 12.625 [4.112 to 21.139] | 6.494 [0.960 to 12.027] | 15.363 [9.078 to 21.647]

15. Secondary Outcome: Change From Baseline in Burden to Others Domain Scores of LupusQoL at Week 52
Description: The LupusQoL questionnaire is a validated questionnaire used to evaluate SLE -specific concepts of SLE as reported by participants. It consists of 34 items in 8 different domains: physical health, emotional health, body image, pain, planning, fatigue, intimate relationship, and burden to others measured on a 5-point scale ranging from 0 (not at all) to 4 (very much). The individual domain scores are transformed to a 0 to 100 scale wherein higher scores indicate better quality of life. Burden to others domain score of LupusQoL had score range from 0 to 100, where higher scores = better quality of life.
Time Frame: Baseline, Week 52
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo | PF-06700841 15 mg | PF-06700841 30 mg | PF-06700841 45 mg
Number analyzed (Participants) | 66 | 36 | 75 | 64
Units on a scale | 12.535 [7.227 to 17.842] | 17.739 [10.412 to 25.065] | 11.560 [6.500 to 16.621] | 18.878 [13.523 to 24.233]

16. Secondary Outcome: Incidence Rate of Severe Flare Event
Description: Incidence rate was defined as the number of new events per 100 person-years.
Time Frame: Week 52
Population: FAS included all participants randomly assigned to study intervention and have received at least 1 dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | Placebo | PF-06700841 15 mg | PF-06700841 30 mg | PF-06700841 45 mg
Number analyzed (Participants) | 96 | 47 | 100 | 97
Events per 100 person-years | 8.32 [3.35 to 17.15] | 6.92 [1.43 to 20.23] | 3.24 [0.67 to 9.46] | 6.95 [2.55 to 15.13]

17. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AE)
Description: An AE was any untoward medical occurrence in a participant who received study intervention without regard to possibility of causal relationship. TEAEs are events from first dose of study intervention to 4 weeks after last dose of study intervention that were absent before treatment or that worsened relative to pre-treatment state. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and all non-SAEs.
Time Frame: Day 1 of dosing up to 4 weeks after last dose of study drug (maximum treatment was up to 52 weeks, follow-up up to 56 weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06700841 15 mg | PF-06700841 30 mg | PF-06700841 45 mg
Number analyzed (Participants) | 100 | 50 | 101 | 99
Participants | 80 | 38 | 88 | 83

18. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study intervention without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: as for outcome 17
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06700841 15 mg | PF-06700841 30 mg | PF-06700841 45 mg
Number analyzed (Participants) | 100 | 50 | 101 | 99
Participants | 8 | 4 | 8 | 9

19. Secondary Outcome: Number of Participants With Adverse Events Leading to Discontinuation From Study
Description: An AE was any untoward medical occurrence in a participant who received study intervention without regard to possibility of causal relationship. In this outcome measure, participants with adverse events leading to discontinuation from study were reported.
Time Frame: as for outcome 17
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06700841 15 mg | PF-06700841 30 mg | PF-06700841 45 mg
Number analyzed (Participants) | 100 | 50 | 101 | 99
Participants | 6 | 2 | 1 | 3

20. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs Abnormalities
Description: Vital signs included blood pressure, pulse rate, respiratory rate, and temperature. Clinical significance in vital signs abnormalities was judged by investigator.
Time Frame: as for outcome 17
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06700841 15 mg | PF-06700841 30 mg | PF-06700841 45 mg
Number analyzed (Participants) | 100 | 50 | 101 | 99
Participants | 0 | 0 | 0 | 0

21. Secondary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: Clinical significance in ECG abnormalities was judged by investigator.
Time Frame: as for outcome 17
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06700841 15 mg | PF-06700841 30 mg | PF-06700841 45 mg
Number analyzed (Participants) | 100 | 50 | 101 | 99
Participants | 0 | 0 | 0 | 0

22. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Hematology (Hemoglobin[hgb], hematocrit, erythrocytes[ery]:<0.8*lower limit of normal[LLN];reticulocytes, reticulocytes/ery:<0.5*LLN,>1.5*upper LN[ULN];ery mean corpuscular volume[EMC], EMC hgb:<0.9*LLN,>1.5*ULN;EMC hgb concentration:<0.9* LLN;platelet:<0.5*LLN;leukocytes[leu]:<0.6*LLN,>1.5*ULN;lymphocytes, lymphocytes/leu, neutrophils, neutrophils/leu:<0.8* LLN,>1.2*ULN;basophils, basophils/leu, eosinophils, eosinophils/leu, monocytes, monocytes/leu:>1.2*ULN;activated partial thromboplastin time[PTT], PTT, prothrombin time:>1.1*ULN);Clinical chemistry (Total/direct/indirect bilirubin, glucose-fasting:>1.5*ULN; aspartate aminotransferase[AT], alanine AT:>3.0*ULN; protein, albumin, HDL cholesterol:<0.8*LLN;urea nitrogen, creatinine, triglyceride, cholesterol:>1.3*ULN;urate, LDL cholesterol:>1.2*ULN;potassium:<0.9*LLN,>1.1*ULN;calcium, bicarbonate:<0.9*LLN;creatine kinase:>2.0*ULN);Urinalysis (pH<4.5;glucose, protein, hgb, ketones, nitrite, leu esterase, granular/hyaline/WBCs casts:>1).
Time Frame: as for outcome 17
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06700841 15 mg | PF-06700841 30 mg | PF-06700841 45 mg
Number analyzed (Participants) | 100 | 50 | 101 | 99
Participants | 96 | 48 | 99 | 97

ADVERSE EVENTS:
Time Frame: Day 1 of dosing up to 4 weeks after last dose of study drug (maximum up to 56 weeks)
Description: Same event may appear as AE and SAE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study.
Arm/Group | Placebo | PF-06700841 15 mg | PF-06700841 30 mg | PF-06700841 45 mg
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/50 | 1/101 | 1/99
Serious Adverse Events (participants affected / at risk) | 8/100 | 4/50 | 8/101 | 9/99
Other Adverse Events (participants affected / at risk) | 47/100 | 19/50 | 53/101 | 47/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=100) | PF-06700841 15 mg (N=50) | PF-06700841 30 mg (N=101) | PF-06700841 45 mg (N=99)
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal strangulation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 2
Cutaneous T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lupus encephalitis (Nervous system disorders) | 0 | 0 | 0 | 1
Thalamic stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Lupus nephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Lupus pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=100) | PF-06700841 15 mg (N=50) | PF-06700841 30 mg (N=101) | PF-06700841 45 mg (N=99)
Diarrhoea (Gastrointestinal disorders) | 5 | 1 | 7 | 6
Nausea (Gastrointestinal disorders) | 5 | 4 | 3 | 7
Vomiting (Gastrointestinal disorders) | 1 | 3 | 4 | 4
Fatigue (General disorders) | 0 | 0 | 6 | 2
COVID-19 (Infections and infestations) | 17 | 9 | 11 | 10
Cystitis (Infections and infestations) | 3 | 3 | 2 | 2
Nasopharyngitis (Infections and infestations) | 7 | 5 | 6 | 8
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 6
Upper respiratory tract infection (Infections and infestations) | 7 | 1 | 11 | 8
Urinary tract infection (Infections and infestations) | 11 | 1 | 10 | 11
Blood creatine phosphokinase increased (Investigations) | 1 | 3 | 1 | 4
Headache (Nervous system disorders) | 5 | 4 | 17 | 9

LIMITATIONS AND CAVEATS:
For the PF-06700841 30 mg, there was a total of 1 death which was reported in both on-treatment and follow-up phases in participant flow section.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT03845517/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-25): https://cdn.clinicaltrials.gov/large-docs/17/NCT03845517/SAP_001.pdf